CLINICAL TRIAL: NCT00897182
Title: Identification of Target Genes for Diagnosis and Prognosis of AML Using a Custom-Design Microarray
Brief Title: Identifying Cancer Genes in in Blood and Bone Marrow Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-20801; CALGB-20801; CDR0000595708 (Registry Identifier: NCI Physician Data Query); NCI-2009-00462 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Microarray Analysis; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bone marrow and/or peripheral blood obtained at diagnosis from AML patients enrolled on CALGB AML treatment studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: This is a CALGB Leukemia Tissue Bank project makes use of tissue from patients who have previously provided their consent. Diagnostic samples from patients enrolled on CALGB AML treatment studies (eg, CALGB 9621, 9710, and 19808) and who have been registered on the companion Leukemia Tissue Bank Protocol CALGB 9665 were used.
  Interventions: Genetic: microarray analysis; Genetic: polymerase chain reaction

INTERVENTIONS:
Genetic: microarray analysis
Genetic: polymerase chain reaction

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify genes related to cancer. It may also help doctors diagnose cancer and predict how patients will respond to treatment.

PURPOSE: This research study is identifying cancer-related genes in blood and/or bone marrow samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify and validate individual genes for diagnosis of three major translocations in acute myeloid leukemia.
* To correlate transcript expression data in the various translocations with age, sex, race, response to treatment, and survival and with other known mutations.

OUTLINE: Blood and/or bone marrow samples previously procured from patients on CALGB-9665 are obtained from the CALGB Leukemia Tissue Bank from patients enrolled on CALGB AML treatment studies. Mononuclear cells are isolated from samples and mRNA is extracted. Gene expression profiles are analyzed via custom mRNA microarray and confirmed by quantitative real-time PCR.

ELIGIBILITY:
* Enrolled on CALGB acute myeloid leukemia (AML) treatment studies AND concurrently enrolled on Leukemia Tissue Bank Protocol CALGB-9665
* Short-term or long-term survivor
* Bone marrow and/or peripheral blood obtained at diagnosis
* Leukemia is one of the following cytogenetic subtypes:

  * t(8;21)
  * t(15;17)
  * inv(16)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with acute myeloid leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2008-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Correlation of increased or decreased expression of same transcripts with disease outcome | baseline
Minimum number of genes that can be used for precise diagnosis of each of the three subtypes of acute myeloid leukemia | baseline
Identification of individual genes that are differentially expressed between the subtypes of AMLs | baseline
Correlation of the patterns of expression of the translocation-specific transcripts with age, sex, race, response to treatment, survival, and with other known mutations | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Janet Rowley, MD, Study Chair — University of Chicago
Locations (2):
- United States (2):
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina